CLINICAL TRIAL: NCT02839759
Title: Interactive Technology for Hearing Aid Education and Acceptance
Brief Title: Hearing Aid Education and Adaptation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthcare Technologies and Methods, LLC (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HTM092016; R44AG045947 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Hearing Loss
Keywords: Hearing loss; Presbycusis; Aging; Teleaudiology
MeSH Terms: conditions — Hearing Loss; Presbycusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELLYHealth Group (Experimental): Subjects will receive the standard of care in hearing aid education and the TELLYHealth intervention for use over an 8 to12-week period and will be followed by their audiologist for 8 to 12 weeks.
  Interventions: Other: TELLYHealth
- Standard of Care Group (No Intervention): Subjects will receive the standard of care in hearing aid education and will be followed by their audiologist for 8 to 12 weeks.

INTERVENTIONS:
Other: TELLYHealth — Educational videos and questions.
  Arms: TELLYHealth Group

SUMMARY:
This RCT will have two arms: A control group that receives the standard of care from audiologists and an experimental group that receives both the standard of care and the at-home use of the TELLYHealth intervention. Subjects in each group will complete questionnaires at enrollment, mid-study and at the end of the study.

DETAILED DESCRIPTION:
HTM will develop the "TELLYHealth (tm) system" that will provide education on hearing aid use and maintenance. HTM will conduct a randomized controlled trial (RCT) to quantify the benefits of TELLYHealth to patients and audiologists including: reductions in hearing handicap, improved knowledge of hearing aid handling, use and communications strategies; and improved audiologist aftercare. The investigators will recruit 80 subjects (half in each group) and each subject will participate in the study for 8-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and reads English fluently
* Has mild (25-40 dB) to severe (70-95 dB) monaural sensorineural hearing loss
* Will be fitted with one or two hearing aids at the time of enrollment
* Owns a standard TV
* Has Internet access at home
* Has sufficient corrected vision to watch videos and read text on the TV and mobile device
* No signs of dementia

Exclusion Criteria:

* Lives with person who has enrolled in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly (HHIE) | 8-12 weeks
  Pre-post changes in the HHIE total scores

SECONDARY OUTCOMES:
Communication Scale for Older Adults (CSOA) | 8-12 weeks
  Pre-post changes in the CSOA communication strategies & attitudes scores

CONTACTS AND LOCATIONS:
Overall Officials: Alan M Letzt, M.S., Principal Investigator — Healthcare Technologies and Methods, LLC
Locations (2):
- United States (2):
  - Clear Sound Audiology, Gainesville, Florida
  - Potomac Audiology, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data on hearing aid education will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: The date will be available approximately May 2025 for one year.
Access Criteria: The criteria will be based on the policies of the selected data repository.